CLINICAL TRIAL: NCT06852105
Title: Compare the Clinical Efficacy of 3% Diquafosol and 0.1% Hyaluronic Acid in Patients with Dry Eye After Trans-PRK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRK2025
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye; Tear Break-Up Time
Keywords: dry eye; Trans-PRK
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Other): dry eye patients after Trans-PRK
  Interventions: Drug: 3% Diquafosol Sodium Eye Drops
- Control group (Other): dry eye patients after Trans-PRK
  Interventions: Drug: 0.1% hyaluronic acid

INTERVENTIONS:
Drug: 3% Diquafosol Sodium Eye Drops — 3% Diquafosol Sodium Eye Drops were instilled into the inferior conjunctival vault of both eyes
  Arms: Study group
Drug: 0.1% hyaluronic acid — 0.1% sodium hyaluronate eye drops were instillation into the inferior conjunctival vault of both eyes
  Arms: Control group

SUMMARY:
The prevalence of refractive ametropia is rising year by year. Refractive surgery has become the main approach for adults to correct refractive ametropia, and postoperative complications have aroused extensive attention from clinicians. Dry eye after refractive surgery is one of the postoperative complications, which is an important cause of affecting the postoperative visual quality and satisfaction of patients. It was reported that 3% diquafosol (DQS) and 0.1% hyaluronic acid (HA) can relieve dry eye symptoms. This study aims to compare the efficacy of 3% DQS and 0.1% HA in treating dry eye after Trans-PRK

DETAILED DESCRIPTION:
The development of corneal refractive surgery is rapid, but the complications are still inevitable; postoperative dry eye is one of them. Dry eye after refractive surgery will affect not only the patient's postoperative satisfaction but also the patient's postoperative visual quality, resulting in blurred vision, not lasting vision, and other problems. The occurrence of postoperative dry eye is mainly due to using anesthetics during operation; corneal nerve injury and cell apoptosis; changes in corneal curvature; postoperative medication, and so on. The patient's bad living habits may aggravate the degree of postoperative dry eye.

Diquafosol sodium is a P2Y2 receptor agonist. P2Y2 receptors are present on conjunctival and corneal epithelial cells, among others, on the ocular surface. When diquafosol sodium is used, it can activate P2Y2 receptors on these cells. This activation triggers the opening of intracellular signaling pathways that stimulate tear secretion. Normal tear secretion is important for corneal nerve repair because tears contain a variety of nutrients and growth factors. In the state of dry eye, the inflammatory factors on the ocular surface increase, and the stability of the tear film decreases. Diquafosol sodium can help to restore the stability of tear film by promoting tear secretion. A stable tear film reduces corneal nerve stimulation by inflammatory factors on the ocular surface. A large area of corneal nerves is injured during Trans-PRK surgery, and no study has shown that diquafosol sodium has a role in nerve recovery after Trans-PRK Hyaluronic acid (HA) lubricates, relieving dry eyes, astringent eyes, and eye fatigue. It can also flush and dilute inflammatory mediators on the ocular surface, reduce tear osmotic pressure, promote ocular surface epithelial healing, and promote ocular surface fibronectin secretion and deposition.

This study aims to compare the efficacy of 3% diquafosol and 0.1% hyaluronic acid in treating dry eye after Trans-PRK. The observation of changes in corneal nerves and immune-inflammatory cells was added, aiming to observe the repair effect of difossol sodium on corneal nerves.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years.
* The refractive status should be maintained at least for more than 2 years, during which the annual increase in myopia should be controlled within 0.50 D.
* Pherical equivalent (SE) ≤-6.00D, astigmatic power≤-2.00D.
* Best corrected vision before surgery≥1.0.
* Patients should stop wearing soft contact lenses for at least 2 weeks and hard contact lenses for at least 4 weeks before surgery.

Postoperative corneal stromal thickness was preserved (280 μm).

Exclusion Criteria:

* Suspected of having keratoconus, a definite diagnosis of keratoconus, or another type of corneal dilatation disease.
* There is active inflammation or symptoms of infection in the eye.
* The thickness of the cornea does not meet the preset cutting depth requirement: the thickness of the central cornea should be greater than 450 μm, and the thickness of the central corneal stroma remaining under the corneal flap should be maintained above 250 μm after the intended cutting (280 μm recommended).
* Dry eye.
* There are serious lesions in the accessory structures of the eye, such as defects or deformations of the eyelids.
* People with uncontrolled systemic connective tissue diseases and autoimmune diseases, such as systemic lupus erythematosus and rheumatoid arthritis.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear break-up time (NITBUT) | day 1, week 1, week 4, week 12 and week 24
  The Keratograph 5M (Oculus, Germany) topographer will assess non-invasive tear breakup time.Three sequential readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.

SECONDARY OUTCOMES:
Conjunctivocorneal staining (CS) | day 1, week 1, week 4, week 12 and week 24
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface
Tear film lipid layer (TFLL) score | day 1, week 1, week 4, week 12 and week 24
  Tear film lipid layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan). The results will be graded as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed
Corneal Sensitivity Score | day 1, week 1, week 4, week 12 and week 24
  Corneal sensitivity score measured with a Cochet-Bonnet esthesiometer (in mm filament length); the measurements will be done 3 times at every assessment session, and the median value will be recorded.
Tear meniscus height (TMH) | day 1, week 1, week 4, week 12 and week 24
  Ear meniscus height using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively, and the median value will be recorded.
Conjunctival hyperemia (RS score): | day 1, week 1, week 4, week 12 and week 24
  Conjunctival hyperemia (RS score) will be assessed by a keratograph image (Oculus, Germany) of 1156 × 873 pixels, with a redness score (RS) ranging from 0.0 (normal) to 4.0 (severe).
Meibomian quality | day 1, week 1, week 4, week 12 and week 24
  Meibomian quality will be assessed under a slit-lamp; eight meibomian glands in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste-like consistency meibum).
Corneal nerves and immune/inflammatory cell change: | 1 week, 12 weeks and 24 weeks after surgery.
  HRT III RCM (Heidelberg Engineering GmbH, Germany) will be used to record corneal nerves and immune/inflammatory cell change. It can accurately scan the cornea from the upper cortex to the inner cortex and other different depth levels and accurately judge the specific level and scope of the lesion. Three representative images of the subbasal nerve plexus and epithelial DCs will be selected for analysis for each eye, considering criteria such as a whole image in the same layer, best focus, and good contrast.
OSDI | day 1, week 1, week 4, week 12 and week 24
  The Ocular Surface Disease Index (OSDI) is a tool used to assess the degree to which ocular surface disease affects a patient's visual function and related symptoms. It is a subjective, patient-self-reported questionnaire. The questionnaire mainly covers three aspects of eye discomfort, including eye pain or discomfort, vision-related dysfunction, and eye irritation symptoms. There are usually 12 questions, and the answer options for each question usually include "none," "mild," "moderate," and "severe," and the corresponding scores are 0, 1, 2, and 3. A range of 0-12 is classified as normal or mild symptoms. A range of 13-22 is classified as moderate symptoms. 23-36 is classified as severe symptoms.
Meibomian gland expressibility | day 1, week 1, week 4, week 12 and week 24
  Meibomian gland expression: five meibomian glands in the middle part were evaluated on a scale of 0-3: 0, all glands expressible; 1, 3-4 glands expressible; 2, 1-2 glands expressible; and 3, no glands expressible.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zaabaar E, Asiamah R, Kyei S, Ankamah S. Myopia control strategies: A systematic review and meta-meta-analysis. Ophthalmic Physiol Opt. 2025 Jan;45(1):160-176. doi: 10.1111/opo.13417. Epub 2024 Nov 12. PMID 39530399
- [Background] Du Y, Di Y, Yang S, Li Y. Analysis of the changes in corneal optical density following small incision lenticule extraction for myopia and related influencing factors. Photodiagnosis Photodyn Ther. 2024 Dec;50:104397. doi: 10.1016/j.pdpdt.2024.104397. Epub 2024 Nov 9. PMID 39528007
- [Background] Mu J, Zhong H, Jiang M, Wang J, Zhang S. Development of a nomogram for predicting myopia risk among school-age children: a case-control study. Ann Med. 2024 Dec;56(1):2331056. doi: 10.1080/07853890.2024.2331056. Epub 2024 Mar 20. PMID 38507901
- [Background] Zhao L, Zhang Y, Duan H, Yang T, Ma B, Zhou Y, Chen J, Chen Y, Qi H. Clinical Characteristic and Tear Film Biomarkers After Myopic FS-LASIK: 1-Year Prospective Follow-up. J Refract Surg. 2024 Aug;40(8):e508-e519. doi: 10.3928/1081597X-20240514-05. Epub 2024 Sep 1. PMID 39120023
- [Background] Hou X, Chen P, Yu N, Luo Y, Wei H, Zhuang J, Yu K. A Comparative and Prospective Study of Corneal Consumption and Corneal Biomechanics After SMILE and FS-LASIK Performed on the Contralateral Eyes With High Myopic Astigmatism. Transl Vis Sci Technol. 2024 Nov 4;13(11):29. doi: 10.1167/tvst.13.11.29. PMID 39576656
- [Background] Yang F, Yang Z, Zhao S, Huang Y. To Investigate the Changes in Corneal Curvature and Its Correlation with Corneal Epithelial Remodeling After Trans-PRK and FS-LASIK. Curr Eye Res. 2024 Oct;49(10):1061-1067. doi: 10.1080/02713683.2024.2361728. Epub 2024 Jun 12. PMID 38867491
- [Background] Su B, Cho P, Vincent SJ, Zheng J, Chen J, Ye C, Wang T, Zhang J, Zhang K, Lu F, Jiang J. Novel Lenslet-ARray-Integrated Spectacle Lenses for Myopia Control: A 1-Year Randomized, Double-Masked, Controlled Trial. Ophthalmology. 2024 Dec;131(12):1389-1397. doi: 10.1016/j.ophtha.2024.07.002. Epub 2024 Jul 6. PMID 38972357